CLINICAL TRIAL: NCT06668597
Title: Evaluation of the Effectiveness of a Brief Motivational Educational Program to Improve Sleep Quality in OSA Patients Through Adherence to CPAP
Brief Title: Educational Motivational Program on Sleep Apnea
Acronym: ME-CA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Eleonora Volpato, Clinical Professor, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ME-CA
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Obstructive Sleep Apnea; Continuous Positive Airway Pressure; Motivational Intervention; Sleep Management; Telemedicine; Psychoeducation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychoeducation Program (Experimental): The experimental group will receive a motivational psychoeducational intervention consisting of four phases: Phase 1 (Pre-adaptation Psychoeducation): The intervention begins with the pulmonologist's decision for home adaptation to CPAP for the patient diagnosed with OSA. The participant will receive necessary materials and an educational video (25 minutes) within two days before the provider's home visit. Phase 2 (Motivational Interview): After the first night of CPAP use, the participant will have a brief motivational interview via phone. Phase 3 (Psychological Support Interview): One week after the provider's intervention, the participant will have a support interview regarding the adaptation process (40 minutes). This first week is a high-risk period for device abandonment. Phase 4 (Monitoring Interview): Two weeks after the provider's intervention, the participant will have a monitoring interview (30 minutes) to check for any difficulties during the adaptation process.
  Interventions: Behavioral: Motivational educational program to improve sleep quality in OSA patients through adherence to CPAP
- Treatment as usual (No Intervention): The patient, following the visit with the pulmonologist specializing in sleep medicine, who has been diagnosed with OSA, will be invited to proceed with the home adaptation process for the CPAP device by the staff.

INTERVENTIONS:
Behavioral: Motivational educational program to improve sleep quality in OSA patients through adherence to CPAP — Phase 1 (Pre-adaptation Psychoeducation): The participant will be shown, within two days prior to the home visit by the provider, which usually takes place within three days of the visit with the pulmonologist, the necessary materials (device, masks, and tubing), along with an educational video on the topic of OSA (duration 25 minutes); Phase 2 (Motivational Interview): Following the first night of titration and use of the CPAP, the participant will be contacted by phone for a brief motivational interview (duration 25 minutes); Phase 3 (Psychological Support Interview): One week after the provider's intervention and the start of the CPAP adaptation period, the participant will be contacted again for a support interview regarding the adaptation process to CPAP (duration 40 minutes). The first week of adaptation is considered a high-risk period for abandonment of device use; Phase 4 (Monitoring Interview): Two weeks after the provider's intervention and the start o
  Arms: Psychoeducation Program

SUMMARY:
The study aims to introduce a motivational intervention for patients with Obstructive Sleep Apnea (OSA) starting CPAP therapy to improve sleep quality and treatment adherence. It will assess average daily CPAP use and compare subjective sleep quality, daytime sleepiness, disease perception, and quality of life between the intervention group and a control group receiving standard care. Inclusion criteria are adults with OSA capable of understanding Italian; exclusion criteria are minors and those already adapted to CPAP. The experimental group will receive a four-phase motivational intervention, while the control group will follow standard CPAP adaptation without additional support.

DETAILED DESCRIPTION:
The study aims to introduce a specific motivational intervention for patients with Obstructive Sleep Apnea (OSA) starting CPAP adaptation, aimed at improving sleep quality and disease management through good adherence to treatment. Additionally, the study will investigate adherence to the proposed treatment in both groups, using average daily use as an adherence indicator, defined as the total hours of CPAP divided by the total number of observation days. Secondary objectives include investigating the effectiveness of the motivational treatment on subjective sleep quality compared to the control group and assessing whether there are statistically significant differences between the clinical practice group (Control Group - GC) and the Experimental Group (GS) in terms of daytime sleepiness (ESS), sleep quality (PSQI), disease perceptions (B-IPQ), and quality of life related to the disease (SF-12). Inclusion criteria are adult patients with OSA (mild, moderate, severe) who are beginning their adaptation process to CPAP and can understand the Italian language. Exclusion criteria include minors, patients already adapted to CPAP, and those unable to understand the Italian language. During the ME-CA study at the Sleep Center, participants will undergo the following procedures to evaluate adaptation to CPAP therapy and its impacts on sleep quality and quality of life. Participants will have an initial evaluation with a pulmonologist in an outpatient setting at the Sleep Center (according to standard clinical practice). They will complete questionnaires to collect socio-demographic data, disease perception, daytime sleepiness, sleep quality, quality of life, and service usability at three different times: at enrollment (T0), one week after the intervention (T1), and three months after the conclusion of the intervention (T2). The adaptation process will follow the assigned protocol (GS or GC); specifically, the Experimental Group will receive a four-phase psychological-motivational intervention in addition to standard CPAP adaptation. Phase 1 (Pre-adaptation psychoeducation): Within two days prior to the home visit by the provider, which typically occurs within three days of the visit with the pulmonologist, participants will be shown an educational video on OSA (25 minutes) and provided with necessary supplies (device, masks, and tubing). Phase 2 (Motivational Interview): After the first night of titration and CPAP use, participants will be contacted for a brief motivational interview (25 minutes). Phase 3 (Psychological Support Interview): One week after the provider's intervention and the start of CPAP adaptation, participants will be contacted for a support interview (40 minutes), as the first week of adaptation is considered a high-risk period for abandoning device use. Phase 4 (Monitoring Interview): Two weeks after the provider's intervention and the beginning of CPAP adaptation, participants will be contacted for a monitoring interview (30 minutes) to ensure no difficulties or issues have arisen during the adaptation process. The frequency and duration of the CPAP adaptation will span a total of 16 days. During this period, participants in the Experimental Group (GS) will engage in four distinct phases, each involving specific meetings or evaluations totaling 120 minutes of participation. These will include psychoeducational sessions, motivational interviews, psychological support, and monitoring. The Control Group (GC), on the other hand, will follow the standard CPAP adaptation pathway without additional meetings or interventions during the initial 15-day adaptation period. Participants in the control group will follow the standard CPAP adaptation pathway. After the visit with the pulmonologist responsible for the Sleep Center, patients in the control group will be offered adaptation to CPAP therapy. They will then be contacted by the provider to arrange a home visit, usually within three days of the visit with the pulmonologist, during which the necessary supplies (device, masks, and tubing) will be provided. Following this, there will be a 15-day adaptation period during which the patient will use the device without further contact with medical staff or the provider. At the end of this period, if the patient has shown adequate adaptability to CPAP therapy, the physician will proceed with the final prescription of the device.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients with OSA (divided, according to the Task Force of the American Academy of Sleep Medicine (Sleep-related breathing disorders in adults: recommendations for syndrome definition and measurement techniques in clinical research. The report of an American Academy of Sleep Medicine Task Force. Sleep. 1999;22(5):667-689) into: Mild OSA with AHI between 5 and 15 Moderate OSA with AHI between 15 and 30 Severe OSA with AHI > 30

* OSA patients who need to begin their home adaptation process to CPAP
* OSA patients who are able to understand the Italian language

Exclusion Criteria:

* Minor patients
* Patients already adapted to CPAP
* Patients unable to understand the Italian language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Brief Illness Perception Questionnaire | At enrollment, one week after the end of the intervention and three months later.
  A self-report questionnaire consisting of 9 items, rated on a 10-point Likert scale, used to assess illness perception, ranging from mild to high.
  All of the items except the causal question are rated using a 0-to-10 response scale. The total score is calculated by summing the scores of all eight items where items 3, 4, and 7 are inversed. The possible range of scores is 0-80. The higher the score, the greater the perceived threat of the illness.
Pittsburgh Sleep Quality Index (PSQI) | At enrollment, one week after the end of the intervention and three months later.
  A self-report questionnaire consisting of 10 items, using a 4-point Likert scale (0-3), used for the subjective assessment of sleep quality over the past month, specifically evaluating dimensions related to sleep efficiency and latency, duration, medication use, the presence of factors disturbing sleep (e.g., pain, heat, etc.), and the impact on quality of life.
  The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Epworth Sleepiness Scale (ESS) | At enrollment, one week after the end of the intervention and three months later.
  A self-report questionnaire consisting of 8 items on a 4-point Likert scale (0-3), used to assess daytime sleepiness in various daily life contexts, such as being a passenger in a car, reading, or attending a theater performance.
  The Epworth sleepiness scale results range from 0 to 24. Results from 0 to 10 show average (normal) daytime sleepiness. A result under 10 may not be cause for concern or it could identify you have trouble sleeping (insomnia). A result from 11 to 24 indicates excessive (abnormal) daytime sleepiness.

SECONDARY OUTCOMES:
Short Form Health Survey - 12 | At enrollment, one week after the end of the intervention and three months later.
  It's the short version of the self-report questionnaire used to assess health-related quality of life and it si compose fog 12 Irene. The scoring of the SF-12 is designed to produce two main scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Each component can have a score ranging from 0 to 100. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Self-Efficacy Measure for Sleep Apnea (SEMSA) | At enrollment and one week after the end of the intervention
  It is a self-report questionnaire consisting of 6 items on a 4-point Likert (1-4) scale, used to assess cognitive factors that may predict patient compliance. Total score consists in the sum of all the item scores (min=6, Max=24). Respondents use a four-point, Likert- type scale ranging from 1 to 4 to indicate their agreement with statements regarding the risks of OSA, their expectations for treatment, and their dedication to CPAP therapy. For each of the instrument's subscales, resulting scores indicate different things. High scores on the perceived risk scale denote greater perceived risks of OSA; high scores on the outcome expectations scale denote more positive beliefs about treatment; high scores on the treatment self-efficacy scale denote a greater willingness to engage in CPAP treatment despite certain obstacles.
System Usability Scale (SUS) | At enrollment, one week after the end of the intervention and three months later.
  It is a self-report questionnaire consisting of 10 items on a 5-point Likert scale (1-5), used to assess the perception of ease of use of the service being utilized.
  SUS is scored on a 10-50, with higher scores indicating a higher perception of ease of use of the service.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Volpato, PhD, Principal Investigator — IRCCS Fondazione Don Gnocchi
Locations (2):
- Italy (2):
  - Don Gnocchi Foundation, Milan, Milan
  - IRCCS Fondazione Don Gnocchi, Milan, MI

IPD SHARING:
Plan to Share IPD: No
The PhD student and psychologist Valentina Poletti will be responsible for the motivational psychological intervention.

REFERENCES:
- [Background] Sampaio R, Pereira MG, Winck JC. Psychological morbidity, illness representations, and quality of life in female and male patients with obstructive sleep apnea syndrome. Psychol Health Med. 2012;17(2):136-49. doi: 10.1080/13548506.2011.579986. Epub 2011 Jul 11. PMID 21745022
- [Background] Poletti V, Battaglia EG, Banfi P, Volpato E. Effectiveness of continuous positive airway pressure therapy on romantic relationships and intimacy among individuals with obstructive sleep apnea: A systematic review and a meta-analysis. J Sleep Res. 2025 Feb;34(1):e14262. doi: 10.1111/jsr.14262. Epub 2024 Jun 24. PMID 38925562
- [Background] Shapiro GK, Shapiro CM. Factors that influence CPAP adherence: an overview. Sleep Breath. 2010 Dec;14(4):323-35. doi: 10.1007/s11325-010-0391-y. Epub 2010 Jul 27. PMID 20661654
- [Background] Lai AYK, Fong DYT, Lam JCM, Weaver TE, Ip MSM. The efficacy of a brief motivational enhancement education program on CPAP adherence in OSA: a randomized controlled trial. Chest. 2014 Sep;146(3):600-610. doi: 10.1378/chest.13-2228. PMID 24810282